CLINICAL TRIAL: NCT04642170
Title: Urodynamic Findings in Patients With Complete and Incomplete Suprasacral Spinal Cord Injury at Different Stages After Injury
Brief Title: Urodynamics of Suprasacral Spinal Cord Injury Patients
Status: Completed | Type: Observational
Sponsor: Second Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Principal Investigator, Junyan Lu, Attending doctor, Second Affiliated Hospital of Wenzhou Medical University
Other Study IDs: SAHoWMU-CR2020-15-212
Record Dates: First submitted 2020-11-14; First posted 2020-11-24 (Actual); Last update posted 2020-11-24 (Actual); Status verified 2020-11

CONDITIONS: Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The medical records of 215 patients with spinal cord injury(SCI) at the Department of Rehabilitation Medicine of the 2nd Affiliated Hospital of Wenzhou Medical University, Wenzhou, China were evaluated between January 1, 2016 and December 20, 2019. According to the inclusion criteria and exclusion criteria, 101 patients were included. The patients were dichotomized into two groups: complete SCI group and incomplete SCI group, based on the American Spinal Injury Association Guidelines Impairment Scale (AIS) .The investigators retrospectively collected records of urodynamic evaluations of this patients and then analyze the urodynamic parameters,including detrusor overactivity (DO), bladder compliance (BC), bladder-filling sensation, maximum cystometric capacity (MCC), detrusor external sphincter dyssynergia (DESD), maximum urinary flow rate (Qmax), detrusor pressure at a maximum urinary flow rate(PdetQmax).

ELIGIBILITY:
Inclusion criteria were:

1. the period of the spinal shock has passed.
2. patients diagnosed with traumatic suprasacral SCI, based on AIS.
3. urodynamic investigations were performed by the same urologist.
4. patients with voiding dysfunction.

Exclusion Criteria:

The patient with voiding dysfunction before the injury were excluded.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Traumatic spinal cord injury patients with voiding dysfunction and had urodynamic examination.
Sampling Method: Non-Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
detrusor overactivity (DO) | 0-365 days after injury
  detrusor overactivity in milliliter,one of the urodynamic parameters
bladder compliance (BC) | 0-365 days after injury
  bladder compliance in ml/cmH2O,one of the urodynamic parameters
bladder-filling sensation | 0-365 days after injury
  bladder-filling sensation,one of the urodynamic parameters

SECONDARY OUTCOMES:
maximum cystometric capacity (MCC) | 0-365 days after injury
  maximum cystometric capacity in milliliter,one of the urodynamic parameters
detrusor external sphincter dyssynergia (DESD) | 0-365 days after injury
  detrusor external sphincter dyssynergia,one of the urodynamic parameters

OTHER OUTCOMES:
maximum urinary flow rate (Qmax) | 0-365 days after injury
  maximum urinary flow rate in milliliter/second,one of the urodynamic parameters
detrusor pressure at a maximum urinary flow rate(PdetQmax) | 0-365 days after injury
  detrusor pressure at a maximum urinary flow rate in cmH2O,one of the urodynamic parameters